CLINICAL TRIAL: NCT04461054
Title: Which Type of Laparoscopic Colectomy, Right or Left, Have Better Postoperative Outcomes for the Patients?
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Leonardo Bustamante-Lopez (Other)
Collaborators: Rodrigo Ambar Pinto (Unknown)
Responsible Party: Sponsor-Investigator, Leonardo Bustamante-Lopez, Colorectal Coordinator of Research at the Sao Paulo University, University of Sao Paulo
Organization: University of Sao Paulo (Other)
Other Study IDs: Colon USP
Record Dates: First submitted 2020-06-28; First posted 2020-07-08 (Actual); Last update posted 2020-07-08 (Actual); Status verified 2020-07

CONDITIONS: Colorectal Disorders
Keywords: colectomy; colorectal; laparoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Laparoscopic surgery decreased the morbidity of colorectal surgery. The two most common surgeries for colorectal cancer are right and left colectomy.

Objective: To compare perioperative morbidity of the right versus left colectomy for cancer, as well as the quality of laparoscopic oncologic resection of both procedures. Methods: Retrospective analysis of prospectively collected data from patients operated at the University of São Paulo School of Medicine, between 2006 and 2016. Postoperative complications were classified with scale within 30 days after surgery. Grade III or greater was considered serious complication. Quality of oncologic resection was assessed by the average number of lymph nodes harvested and surgical margins.

DETAILED DESCRIPTION:
Laparoscopic surgery decreased the morbidity of colorectal surgery. The two most common surgeries for colorectal cancer are right and left colectomy.

This retrospective analysis of prospectively collected data from patients operated at the University of São Paulo School of Medicine, between 2006 and 2016. Postoperative complications were classified by scale within 30 days after surgery. There were 332 patients operated.

ELIGIBILITY:
Inclusion Criteria: patients who underwent laparoscopic right or left elective colectomy for colon adenocarcinoma.

Exclusion Criteria: Patients who underwent total colectomy

* Resections that included the rectum
* Exclusive transverse resections
* Multivisceral resections

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: colon adenocarcinoma
Sampling Method: Non-Probability Sample
Enrollment: 332 (Estimated)
Dates: Start 2020-01-02 (Actual); Primary Completion 2020-09-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative complications | 30 days
  Complications

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo A Pinto, MD, PhD, Principal Investigator — University of Sao Paulo
Locations (1):
- Medicine School, Sao Paulo University, São Paulo, Brazil